CLINICAL TRIAL: NCT02834520
Title: Expression of miRNA-138 and Cyclin D1 in Oral Lichen Planus (A Study Utilizing Immunohistochemistry and Real-time Polymerase Chain Reaction)
Brief Title: Expression of miRNa-138 and Cyclin D1 in Oral Mucosa of Patients With Oral Lichen Planus
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of Oral Medicine and Periodontology, Cairo University
Other Study IDs: MiRNA-138_cyclin D1_OLP
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — oral mucosa tissue specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- oral lichen planus: 30 patients suffering from reticular, erosive and atrophic oral lichen planus
- control subjects: 30 individuals age, gender and periodontal status matched with oral lichen planus patients and not suffering from any oral mucosal lesions or periodontal disease.

SUMMARY:
60 individuals were subdivided into 2 groups, 30 patients with oral lichen planus, 30 control individuals. Expression of miRNA-138 and cyclin D1 were evaluated in oral mucosa utilizing Quantitative real-time polymerase chain reaction and immunohistochemistry.

DETAILED DESCRIPTION:
60 individuals were subdivided into 3 groups, into 2 groups, 30 patients with oral lichen planus, 30 control individuals having age, gender and periodontal status matched with both patients groups acting as a control group. Relative gene expression of miRNA-138 was estimated using Quantitative real-time polymerase chain reaction technique in oral mucosa of both oral lichen planus patients and control subjects. Sub grouping of oral lichen planus patients were performed into reticular, atrophic and erosive groups (n=10 each). Cyclin D1 gene expression was estimated using Quantitative real-time polymerase chain reaction technique and Cyclin D1 protein level was estimated using immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral lichen planus.

Exclusion Criteria:

* any systemic disease other than oral lichen planus.
* smokers.
* pregnant females.
* periodontal diseases.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 individuals were subdivided into 2 groups, 30 patients suffering from oral lichen planus and 30 individuals having age, gender and periodontal status matched with both patients groups acting as a control group.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
expression of miRNA-138 | 1 day
  expression of miRNA-138 in oral mucosa of patients with oral lichen planus

SECONDARY OUTCOMES:
gene expression of cyclin D1 | 1 day
  gene expression of cyclin D1 in oral mucosa of patients with oral lichen planus
protein expression of cyclin D1 | 1 day
  protein expression of cyclin D1 in oral mucosa of patients with oral lichen planus

CONTACTS AND LOCATIONS:
Overall Officials: Noha Ghallab, MD, Principal Investigator — Associate Professor of periodontology and Oral Medicine faulty of oral an

REFERENCES:
- [Result] Jiang L, Liu X, Kolokythas A, Yu J, Wang A, Heidbreder CE, Shi F, Zhou X. Downregulation of the Rho GTPase signaling pathway is involved in the microRNA-138-mediated inhibition of cell migration and invasion in tongue squamous cell carcinoma. Int J Cancer. 2010 Aug 1;127(3):505-12. doi: 10.1002/ijc.25320. PMID 20232393
- [Result] Liu X, Jiang L, Wang A, Yu J, Shi F, Zhou X. MicroRNA-138 suppresses invasion and promotes apoptosis in head and neck squamous cell carcinoma cell lines. Cancer Lett. 2009 Dec 28;286(2):217-22. doi: 10.1016/j.canlet.2009.05.030. Epub 2009 Jun 21. PMID 19540661
- [Result] Jin Y, Chen D, Cabay RJ, Wang A, Crowe DL, Zhou X. Role of microRNA-138 as a potential tumor suppressor in head and neck squamous cell carcinoma. Int Rev Cell Mol Biol. 2013;303:357-85. doi: 10.1016/B978-0-12-407697-6.00009-X. PMID 23445815
- [Result] Liu X, Lv XB, Wang XP, Sang Y, Xu S, Hu K, Wu M, Liang Y, Liu P, Tang J, Lu WH, Feng QS, Chen LZ, Qian CN, Bei JX, Kang T, Zeng YX. MiR-138 suppressed nasopharyngeal carcinoma growth and tumorigenesis by targeting the CCND1 oncogene. Cell Cycle. 2012 Jul 1;11(13):2495-506. doi: 10.4161/cc.20898. Epub 2012 Jul 1. PMID 22739938
- [Result] Yao X, Yin C, Shen LJ, Xie SM. [Expressions of NF--kappaBp65, TRAF2, cyclinD1 and their association with cell apoptosis in oral lichen planus]. Nan Fang Yi Ke Da Xue Xue Bao. 2007 Nov;27(11):1657-60. Chinese. PMID 18024283
- [Result] Hirota M, Ito T, Okudela K, Kawabe R, Yazawa T, Hayashi H, Nakatani Y, Fujita K, Kitamura H. Cell proliferation activity and the expression of cell cycle regulatory proteins in oral lichen planus. J Oral Pathol Med. 2002 Apr;31(4):204-12. doi: 10.1034/j.1600-0714.2002.310403.x. PMID 12076323